CLINICAL TRIAL: NCT02747056
Title: Study of the Personal Identity in Adults With Autism Spectrum Disorder Without Intellectual Deficiency
Acronym: TSASDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6282
Record Dates: First submitted 2016-03-07; First posted 2016-04-21 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Autism spectrum disorder studyA part1 (Experimental): The subjects will perform clinical, psychological and neuropsychological assessment. the subjects will do 3 tests about executive functions. Finally, the participants will complete 3 questionnaires about autism and 3 questionnaires about the self concept.
- Autism spectrum disorder studyA part2 (Experimental): The subjects will perform Autobiographical memories Assessment. The subjects will tell autobiographical memories freely first and secondly by answering focused questions to specify the characteristics of subjects' memories
  Interventions: Other: Autobiographical memories Assessment
- Control adults Study A, part 1 (Other): The subjects will perform clinical, psychological and neuropsychological assessment. The subjects will do 3 tests about executive functions. The participants will complete 3 questionnaires about autism and 3 questionnaires about the self concept.
  Interventions: Other: clinical, psychological and neuropsychological assessment
- Control adults Study A, part 2 (Other): The subjects will perform Autobiographical memories Assessment. The subjects will tell autobiographical memories freely first and secondly by answering focused questions to specify the characteristics of subjects' memories
  Interventions: Other: Autobiographical memories Assessment
- Autism spectrum disorder Study B, part 1 (Experimental): The subjects will perform clinical, psychological and neuropsychological assessment. The subjects will do 3 tests about executive functions. The participants will complete 3 questionnaires about autism and 3 questionnaires about the self concept.
  Interventions: Other: clinical, psychological and neuropsychological assessment
- Autism spectrum disorder Study B, part 2 (Experimental): The subjects will perform Autobiographical memories assessment characteristics. The subjects will say the self statements which define them. Then, the participants will have to tell and specify the characteristics of the autobiographical memories linked to the self statements.
  Interventions: Other: Autobiographical memories assessment characteristics
- Control adults, Study B part 1 (Other): The subjects will perform clinical, psychological and neuropsychological assessment.The subjects will do 3 tests about executive functions. Finally, the participants will complete 3 questionnaires about autism and 3 questionnaires about the self concept.
  Interventions: Other: clinical, psychological and neuropsychological assessment
- Control adults, Study B part 2 (Other): The subjects will perform Autobiographical memories assessment characteristics. The subjects will say the self statements which define them. Then, the participants will have to tell and specify the characteristics of the autobiographical memories linked to the self statements
  Interventions: Other: Autobiographical memories assessment characteristics

INTERVENTIONS:
Other: clinical, psychological and neuropsychological assessment — the subjects will do 3 tests about executive functions, complete 3 questionnaires about autism and 3 questionnaires about the self concept
  Arms: Autism spectrum disorder Study B, part 1; Control adults Study A, part 1; Control adults, Study B part 1
Other: Autobiographical memories Assessment — The investigators will ask subjects to tell autobiographical memories freely first and, secondly, to specify participants'characteristics by answering focused questions.
  Arms: Autism spectrum disorder studyA part2; Control adults Study A, part 2
Other: Autobiographical memories assessment characteristics — During the second time point, the investigators will ask subjects to say the self statements which define them. Then, subjects will have to tell and to specify the characteristics of the autobiographical memories linked to these self statements.
  Arms: Autism spectrum disorder Study B, part 2; Control adults, Study B part 2

SUMMARY:
The research aims at clarifying the impact of autism on personal identity in adulthood. Two studies will be made in order to compare adults with autistic spectrum disorders without intellectual deficiency and controls. In the first study (Study A), the investigators will ask subjects to tell autobiographical memories and to specify their characteristics by answering focused questions. In the second study (Study B), the investigators will ask subjects to say the self statements which define them. Then, subjects will have to tell and to specify the characteristics of the autobiographical memories linked to these self statements.

DETAILED DESCRIPTION:
Introduction:

Autism associates impairments in social relationships and specific competencies linked to restricted interests. These interests usually focus on mathematics, drawings or foreign language learning and are very significant in the autobiographies of persons with autism without intellectual deficiency. It's seem to be a basement of their self-identity. The personal identity relies on both the self representations and the sense of self. This sense of self supports the self continuity through time which links the present feelings, the autobiographical memories and the future personals projects. The personal identity depends on the memory of life events called "autobiographical memory."

Objectives:

The research aims at clarifying the impact of autism on personal identity in adulthood. Two studies will be made in order to compare adults with autistic spectrum disorders without intellectual deficiency and controls. In the first study (Study A), the investigators will ask subjects to tell autobiographical memories and to specify their characteristics by answering focused questions. In the second study (Study B), the investigators will ask subjects to say the self statements which define them. Then, subjects will have to tell and to specify the characteristics of the autobiographical memories linked to these self statements.

Expected Results:

The first study will inform the investigators on the sense of self and self continuity through time. The investigators predict that it would be difficult for subjects with autism spectrum disorders to give details of their life events. The focused questions should make easier the recollection of the memories. The investigators hypothesize that the memories linked to the typically autistic restricted interests would be more detailed.

The second study will inform the investigators on the memories linked to self representations. The investigators predict that these memories would be, in autism, less detailed and less important for identity. The investigators also hypothesize that the memories linked to the restricted interests would be more detailed and important for the self.

Autobiographical memory and socialization are deeply interconnected. So, the investigators think that this research will help them to elaborate news therapies focused on autobiographical memory improvement. Finally, the investigators want to reduce the social disability in autism.

ELIGIBILITY:
Study A & B, Adults with autism spectrum disorders without intellectual deficiency

Inclusion criteria:

* adults with autism spectrum disorders
* 18 to 65 years old

Exclusion criteria:

* treatment with benzodiazepines

Study A & B, control adults

Inclusion criteria:

* healthy volunteers
* 18 to 65 years old

Exclusion criteria:

* psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
The number of details in the memory (A)/The specificity of the memory (B) | The number of details or the specificity of the memory is assessed from 1 day to 3 months after the inclusion/baseline
  study A:The number of details is the total number of perceptual/sensory, temporal, contextual, emotional and cognitive details found in the memory after spontaneous recall first. Secondly, the investigators will ask subjects to clarify the five characteristics of the details presented upper and retrieval should be make easier with specific cueing.
  Study B:The specificity measures how the memory is focused on specific date, space, context, emotions, thoughts and feelings. The specificity of the memories is deeply linked to the self .

SECONDARY OUTCOMES:
Study A and B: Autistic symptoms questionnaire 1 | the Autistic symptoms will be assessed during the initiation/baseline visit at V1
  Autistic symptoms are assessed through the Ritvo's Autism Asperger Diagnostic Scale. A numerical value will be obtained for this questionnaire.
Study A and B: Autistic symptoms questionnaire 2 | the Autistic symptoms will be assessed during the initiation/baseline visit at V1
  Autistic symptoms are assessed through the Empathy Quotient. A numerical value will be obtained for this questionnaire.
Study A and B: Autistic symptoms questionnaire 3 | the Autistic symptoms will be assessed during the initiation/baseline visit at V1
  Autistic symptoms are assessed through the Autistic Quotient. A numerical value will be obtained for this questionnaire.
Study A and B:Executives functions, test 1 | Executives functions will be assessed during the initiation/baseline visit (V1)
  Executive functions are measured through test: the Trail Making Test A & B, The test will provide value in seconds. This executive functions are known to be impaired in autism spectrum disorder and to be involved in autobiographical memory.
Study Aand B:Executives functions test 2 | Executives functions will be assessed during the initiation/baseline visit (V1)
  Executive functions are measured through test: The Hayling test . The tests will provide value in seconds. This executive functions are known to be impaired in autism spectrum disorder and to be involved in autobiographical memory.
Study A and B:Executives functions test 3 | Executives functions will be assessed during the initiation/baseline visit (V1)
  Executive functions are measured through test: The phonologic verbal fluency tasks. The test will give numerical value. These executive functions are known to be impaired in autism spectrum disorder and to be involved in autobiographical memory.
Study A and B: The self concept, questionnaire 1 | self-concept will be assessed during the initiation/baseline visit (V1)
  The self-concept is measured through the questionnaire like the Thinking About Life Experiences (TALE) scale. This test measure how the self is updated and adaptable. A numerical value will be obtained for the questionnaire.
Study A and B: The self concept, questionnaire 2 | self-concept will be assessed during the initiation/baseline visit (V1)
  The self-concept is measured through the questionnaire like: The Self Concept Clarity Scale. This test measure how the self is updated and adaptable. A numerical value will be obtained for the questionnaire.
Study A and B: The self concept, questionnaire 3 | self-concept will be assessed during the initiation/baseline visit (V1)
  The self-concept is measured through the questionnaire like : The Rosenberg self-esteem test. This test measure how the self is updated and adaptable. A numerical value will be obtained for the questionnaire.
Study A: the number of remember/ know/ guess responses, the perspective in recollection and the subjective temporal distance in the memory | This outcome will be assessed on the follow up visit (V2) either one day after the inclusion visit (V1) or within 3 months after V1
  The number or remember, know, guess responses gives information about the subjective state of conscious awareness during the recall of the memory. This subjective state goes from complete conscious recollection with reliving of thoughts, perceptions, and feelings at the date of the event to a vague impression.
  The perspective in recollection could be an actor perspective or an observer perspective. In the actor perspective, the recollection is in a first-person point of view. The person remembering relives the event through her own eyes. In the observer perspective, the recollection is in a third-person point of view. The person remembering sees the scene of the memory as the spectator of herself.
  The subjective temporal distance is the subjective perception of the temporal distance between the present and the event of the memory. The investigators will ask subjects if they feel this event close or distant on a seven point scale.
Study B:The importance for the self of the memory test1 | This outcome will be assessed on the follow up visit (V2) either one day after the inclusion visit (V1) or within 3 months after V1Description
  The importance for the self of the memory is assessed by distinctiveness. The distinctiveness criteria of the memory is established by Conway. These criteria require participants to specify in what extent these memories have had a personal significance, were discriminatory, consistent and are frequently recalled. A numerical value will be obtained for this criteria.
Study B:The importance for the self of the memory test 2 | this outcome will be assessed on the follow up visit (V2) either one day after the inclusion visit (V1) or within 3 months after V1Description
  The importance for the self of the memory is assessed by emotional intensity. The emotional intensity will be measured with the PANAS scale. The investigator will ask the participants to rate the emotional intensity of their memory based on 4 positive affect (determined, enthusiastic, proud and strong) and 4 negative affect (frightened, ashamed, guilty and disappointed). No value is obtained.
Study B:The importance for the self of the memory test 3 | this outcome will be assessed on the follow up visit (V2) either one day after the inclusion visit (V1) or within 3 months after V1Description
  The importance for the self of the memory is assessed by the active or passive position . An active position will refer to a memory in which the subject plays a key role in the progression of the event. A passive position will refer to a memory where the participant undergoes an event where he did not play a determining role.
Study B:The importance for the self of the memory test 4 | this outcome will be assessed on the follow up visit (V2) either one day after the inclusion visit (V1) or within 3 months after V1Description
  The importance for the self of the memory is assessed by the emotional valence of memory. The emotional valence of memory will be etheir positive, negative or neutral.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marie DANION, Prof, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coutelle R, Goltzene MA, Bizet E, Schoenberger M, Berna F, Danion JM. Self-concept Clarity and Autobiographical Memory Functions in Adults with Autism Spectrum Disorder Without Intellectual Deficiency. J Autism Dev Disord. 2020 Nov;50(11):3874-3882. doi: 10.1007/s10803-020-04447-x. PMID 32146597